CLINICAL TRIAL: NCT02771327
Title: Phase 4, Randomized, Controlled Trial on the Efficacy as Prophylaxis of Postoperative Respiratory Complications and Safety of Continuous Positive Airways Pressure (CPAP) Applied Throughout Boussignac Mask During the Immediate Postoperative Period of Patients Undergoing Lung Resection
Brief Title: Use of a Pressurized Face Mask for Preventing Respiratory Complications After Chest Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIBHGM-ECNC010-2010
Record Dates: First submitted 2016-04-04; First posted 2016-05-13 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Lung Resection
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP plus gas (Experimental): Treatment with Boussingnac valve CPAP during 6 hour, starting immediately after weaning
  Interventions: Device: CPAP plus Gas
- Usual treatment(ventimask plus gas) (Active Comparator): ventimask
  Interventions: Device: ventimask plus gas

INTERVENTIONS:
Device: CPAP plus Gas
  Arms: CPAP plus gas
Device: ventimask plus gas
  Arms: Usual treatment(ventimask plus gas)

SUMMARY:
Evaluation of efficacy and safety from 6hours of 7 cmH2O CPAP after weaning in patients undergoing lung resection, on the prevention of atelectasis / pneumonia and gas exchange improve.

DETAILED DESCRIPTION:
Multicenter randomized clinical trial. 460 patients randomly assigned to treatment and control groups will be studied. The main variables are the frequency of atelectasis or pneumonia, defined by clinical and radiological criteria, the FiO2/PaO2 ratio, 7 and 24 h after weaning, and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing thoracic surgery including resection of lung parenchyma.
* To have given signed consent to enter in the study.

Exclusion Criteria:

Weaning in the first 4h after the intervention end.

* Suspected bronchopleural fistula at the admission to the surgical ICU.
* Patients with facial problems or a history of intolerance to CPAP masks.
* Having significant bullous emphysema defined as the presence of more than 5 contiguous bullae <2cm or the existence of a pulmonary bulla> 2 cm or dystrophy bullosa, not in the area to dry and having had a previous pneumothorax.
* Known Obstructive Apnea Hypopnea syndrome known or some form of noninvasive ventilation prescribed.
* Immunocompromised patients, or having used an immunosuppressor drug at least one month prior to surgery with potential (except corticosteroids administered by inhalation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2014-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Frequency of atelectasis- Pneumonia, and other postoperative complications, | 1 week after the surgical intervention

SECONDARY OUTCOMES:
Gas exchange ( Pa/FiO2) | 1 week after the surgical intervention
Hospital stay comparison between arms | from the surgical intervention date to hospital discharge date up to 1month

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hopsital universitario La Princesa, Madrid, Madrid
  - HGU Gregorio Marañón, Madrid, Madrid
  - H. Ramón y Cajal, Madrid, Madrid
  - HU 12 de octubre, Madrid, Madrid